CLINICAL TRIAL: NCT03690232
Title: Comparison of the Clinical Efficacy of Intraarticular Glucose Versus Hyaluronic Acid Injection for Knee Osteoarthrosis
Brief Title: Intraarticular Glucose Versus Hyaluronic Acid Injection for Knee Osteoarthrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-01-014C
Record Dates: First submitted 2018-09-09; First posted 2018-10-01 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: The study in the first year is a prospective, randomized controlled, double-blind study. The enrolled patients were randomly divided into two groups: the intraarticular glucose group and the intraarticular HA group.
Who Masked: Participant, Outcomes Assessor
Masking Description: outcomes assessor and participant do not know the treatment patient received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucose group (Experimental): The glucose group underwent 3 sessions of 6cc 25% glucose injection with a 2-week interval between each treatment
  Interventions: Drug: glucose water
- hyaluronic acid group (Active Comparator): The HA group was administered intra-articular HA ((Hyruan Plus® , average MW 3000 kD; LG Life Sciences Ltd, Korea)) for sessions with a 1-week interval between each treatment.
  Interventions: Drug: hyaluronic aicd

INTERVENTIONS:
Drug: glucose water — 3 sessions of 6cc 25% glucose injection with a 2-week interval
  Arms: Glucose group
Drug: hyaluronic aicd — intra-articular HA ((Hyruan Plus® , average MW 3000 kD; LG Life Sciences Ltd, Korea)) for sessions with a 1-week interval between each treatment
  Other Names: Hyruan
  Arms: hyaluronic acid group

SUMMARY:
The study is a prospective, randomized controlled, double-blind study. The enrolled patients were randomly divided into two groups: the intraarticular glucose group and the intraarticular HA group.

DETAILED DESCRIPTION:
The glucose group underwent 3 sessions of 6cc 25% glucose injection with a 2-week interval between each treatment. The HA group was administered intra-articular HA ((Hyruan PlusR, average MW 3000 kD; LG Life Sciences Ltd, Korea)) for sessions with a 1-week interval between each treatment. The results were measured with the visual analogue scale (VAS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), and Lequesne index. A baseline for each test was measured before treatment and then the effects of the treatments were measured by each test at 6 and 12 weeks after treatment

ELIGIBILITY:
Inclusion Criteria:

1. people aged 45 years or more;
2. subjects diagnosed with knee OA according to the clinical criteria of the American College of Rheumatology
3. subjects diagnosed with grade II or III OA during radiological examination as defined by the radiological classification of Kellgren and Lawrence (K-L) scale for knee OA
4. subjects with tenderness in the medial tibial plateau area

Exclusion Criteria:

1. . subjects having other illnesses of neurologic diseases, cardiac disorders, hemodynamically unstable systems, or physical functions;
2. . Inflammatory arthritis or subjects with acute knee arthritis
3. . subjects who have received intraarticular injection on the affected knee within the past 3 months.
4. . subjects with previous medical histories involving the affected knee such as surgeries, cancer and maligament tumors.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-10-08 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 12 weeks
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales

SECONDARY OUTCOMES:
Lequesne index | 0,6,12 weeks
  The Lequesne Index is a 10-question survey given to patients with osteoarthritis of the knee. It has five questions pertaining to pain or discomfort, 1 question dealing with maximum distance walked, and four questions about activities of daily living
visual analogue scale (VAS) | 0,6,12 weeks
  pain intensity was measured by VAS from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Jia chi Wang, MD, Study Director — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No